CLINICAL TRIAL: NCT04472624
Title: Short Term Induction of Ketosis in PKD
Acronym: RESET-PKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Roman Müller, Department II of Internal Medicine, University of Cologne
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20-1040
Record Dates: First submitted 2020-06-09; First posted 2020-07-15 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: ADPKD
Keywords: ADPKD; dietary intervention; ketosis; fasting; ketogenic diet
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Ketosis; Fasting | interventions — Angptl4 protein, mouse; Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting arm (Experimental): Participants will be fasting during 72 hours
  Interventions: Other: Fasting
- Diet arm (Experimental): Participants will be using ketogenic diet for 14 days
  Interventions: Other: Ketogenic diet

INTERVENTIONS:
Other: Fasting — Acute fasting for 72 hours
  Arms: Fasting arm
Other: Ketogenic diet — Intake of a ketogenic diet for 14 days
  Arms: Diet arm

SUMMARY:
Recently, it has been shown that ketose-inducing dietary interventions slow disease progression in animal models of polycystic kidney disease (PKD), even when the state of ketosis is only induced for a short period of time. The present study aims to investigate the effects of short term ketosis on total kidney volume (TKV) (and other parameters) in 10 ADPKD-patients with rapidly progressive disease.

DETAILED DESCRIPTION:
Recently, dietary models inducing ketosis have been shown to inhibit disease progression in animal models of PKD. Those beneficial dietary models included time-restricted feeding (TRF) without caloric reduction, ad libitum administered ketogenic diet (KD) and acute short-term fasting in mouse, rat and feline models of PKD.

In a PKD rat model, TRF without caloric reduction resulted in a strong inhibition of mTOR signaling, proliferation and fibrosis in the affected kidneys. The adminstration of an ad libitum fed KD led to similar results. In rat, mouse and feline models of PKD, acute fasting led to a significant reduction of cyst volume. Therefore, cystic cells seem to be metabolically inflexible and exhibit an altered metabolism characterized by increased glycolysis and, amongst others, defective fatty acid oxidation, similar to the Warburg effect in cancer. (Torres, Kruger et al. 2019)

While those beneficial observations were made in mouse, rat and feline models of PKD, the effects of a ketogenic diet in human ADPKD patients have not been investigated yet, even though the adminstration of ketogenic diets is used as a treatment for epilepsy in children since the 1920s and fasting is one of the oldest medical procedures.

Therefore, the aim of the present study is to investigate the effects of a short-period ketonic state in 10 ADPKD patients with fast progressive disease.

10 ADPKD-patients (aged 18-60 years, CKD G 1-3a) will be enrolled after giving informed consent. These 10 subjects will go through four trial-related visits. During these visits, physical examinations will be performed, blood will be drawn, urine will be collected and ketone body measurements in breath, blood and urine will be carried out. Each study visit includes an abdominal MRI-scan. Between visit 1 and visit 2, patients will eat their regular carbohydrate-rich diet. After visit 2, a ketonic state will be induced in those patients. Patients can choose whether the ketonic state will be induced by acute fasting for 72 hours (under sufficient water consumption and salt substitution) or by eating a KD for 14 days. Study visit 3 will take place within 72 hours after finishing the dietary intervention. After study visit 3, patients will restart eating their regular diet. Study visit 4 will provide follow-up data 3-6 weeks after the dietary intervention.

After study completion, the relative difference of TKV measured by MRI-based volumetry of the kidneys immediately before and immediately after the ketonic state, will be compared to TKV growth/decline while eating a regular carbohydrate-rich diet.

In general, patients are counselled in our outpatient department as part of "The German AD(H)PKD Registry" (more than 700 patients enrolled). As from those patients, clinical data, laboratory data and imaging studies are present, identification and recruitment of patients with fast rapidly progressing disease will be facilitated. Also, the investigators are closely liaised with the German self-help group PKDCure (PKD Familiaere Zystennieren e.V.), which is dedicated to ADPKD-linked research. This will facilitate recruitment of patients even more.

Data obtained from the study visits will be collected. The parameters listed below constitute the core data set, additional parameters can be included if considered essential.

Registered patients will be provided with diaries for the documentation of feeling of hunger, problems and discomforts as well as acetoacetate concentrations in breath. Patients are also provided with a portable breath-analyzer to measure acetoacetate concentrations in breath in between study visits. Study diaries are collected on Visit 4.

Data capture will be performed at each study visit after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female ADPKD-patients (diagnosed by genetics / typical MRI / ultrasound)
* With evidence of fast progression, at least one of the following criteria

  1. Mayo Class 1C-1E
  2. Truncating PKD1-mutation
  3. Hypertension < 35 years
  4. Urological complications < 35 years
  5. ≥ 1 first class or second class family member with need of renal replacement therapy < 60 years
  6. eGFR loss > 2,5 ml/min/1,73m2 per year
  7. PROPKD-Score > 6
* Age ≥ 18 and ≤ 60 years
* CKD stage 1-3a according to eGFR
* Signed written informed consent

Exclusion Criteria:

* Currently under tolvaptan
* BMI < 18 or > 35
* Diabetes mellitus (Type I, Type II, MODY, LADA)
* Active alcoholism
* Vegan or vegetarian lifestyle
* Inability to sign or understand written informed consent
* Anamnestically known circumstances which forbid the induction of a ketonic state by ketogenic diet or acute fasting (Liver damage (AST/ALT > 3x upper limit of normal, alkaline phosphatase > 6x upper limit of normal , Bilirubin ≥ 3 mg/dl), Diabetes mellitus, Pyruvate carboxylase deficiency, defects of gluconeogenesis, defects of ketolysis / ketogenesis, hyperinsulinism, defects of fatty acid oxidation )
* Allergies or food intolerance against components of a ketogenic diet
* Eating disorders (Anorexia nervosa / Bulimia)
* Participation in a weight loss program (e.g. Optifast) or intake of medication to promote weight loss within the last six months
* Ketogenic Diet > 1 month within the last 12 months
* Chronic renal replacement therapy
* Previous history of kidney transplantation
* Uncontrolled local or systemic infection (according to clinical assessment)
* Simultaneous participation in other interventional studies
* Pregnant or breastfeeding women
* Persons who are dependent of or employed by the study investigators
* Contraindications against MRI examinations (stents, pacemakers or other metal inserts, claustrophobia)
* Persons living in an establishment by court order or official instructions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Relative difference of TKV immediately before and after the ketonic state | Visit 2: 2-4 Weeks after enrolment; Visit 3: 3 - 21 days after Visit 2
  MRI-based kidney volumetry at study visit 2 and study visit 3

SECONDARY OUTCOMES:
Absolute and relative difference of TKV | Baseline visit (V1) and final study visit (V4) after at maximum 95 days
  assessed by MRI-based volumetry at all study visits
Absolute and relative difference of height-adjusted total kidney volume (htTKV) | Baseline visit (V1) and final study visit (V4) after at maximum 95 days
  assessed by MRI-based volumetry at all study visits
Absolute and relative difference of total liver volume (TLV) | Baseline visit (V1) and final study visit (V4) after at maximum 95 days
  assessed by MRI-based volumetry at all study visits
Absolute and relative difference of cystic burden of kidneys and liver | Baseline visit (V1) and final study visit (V4) after at maximum 95 days
  assessed by MRI at all study visits
Absolute and relative change of Renal Function Panel | Baseline visit (V1), study visit 2 (V2): 2-4 Weeks after enrolment; Visit 3: 3 - 21 days after Visit 2, and final study visit (V4) after at maximum 95 days
  Measurement of creatinine, urea and uric acid in blood and urine samples (measurement unit mg/dl)
Absolute and relative change of electrolytes and minerals | Baseline visit (V1), study visit 2 (V2): 2-4 Weeks after enrolment; Visit 3: 3 - 21 days after Visit 2, and final study visit (V4) after at maximum 95 days
  Measurement of electrolyte and minerals (sodium, natrium, potassium, magnesium, chloride, phosphate) in blood (measurement unit mmol/L) and urine samples (measurement unit mmol/24h)
Absolute and relative change of albumin | Baseline visit (V1), study visit 2 (V2): 2-4 Weeks after enrolment; Visit 3: 3 - 21 days after Visit 2, and final study visit (V4) after at maximum 95 days
  Measurement in blood and urine samples
Absolute and relative change of glucose | Baseline visit (V1), study visit 2 (V2): 2-4 Weeks after enrolment; Visit 3: 3 - 21 days after Visit 2, and final study visit (V4) after at maximum 95 days
  Measurement in blood and urine samples
Absolute and relative change of Hepatic Function Panel | Baseline visit (V1), study visit 2 (V2): 2-4 Weeks after enrolment; Visit 3: 3 - 21 days after Visit 2, and final study visit (V4) after at maximum 95 days
  Measurement of Alanine aminotransferase(ALT), Aspartate Aminotransferase (ASP), Alkaline Phosphatase (ALP), gamma-glutamyl transferase (GGT) and Lactate Dehydrogenase (LD) in blood samples (measurement unit U/L)
Absolute and relative change of bilirubin | Baseline visit (V1), study visit 2 (V2): 2-4 Weeks after enrolment; Visit 3: 3 - 21 days after Visit 2, and final study visit (V4) after at maximum 95 days
  Measurement in blood samples
Absolute and relative change of lipid panel | Baseline visit (V1), study visit 2 (V2): 2-4 Weeks after enrolment; Visit 3: 3 - 21 days after Visit 2, and final study visit (V4) after at maximum 95 days
  Measurement of high density lipoprotein (HDL), low density lipoprotein (LDL), total cholesterol, triglycerides and lipoprotein(a) in blood samples
Absolute and relative change of inflammatory parameters | Baseline visit (V1), study visit 2 (V2): 2-4 Weeks after enrolment; Visit 3: 3 - 21 days after Visit 2, and final study visit (V4) after at maximum 95 days
  Measurement of c-reactive protein (CRP) and high sensitivity c-reactive protein (hsCRP) in blood samples ( measurement unit mg/L)
Absolute and relative change in blood count | Baseline visit (V1), study visit 2 (V2): 2-4 Weeks after enrolment; Visit 3: 3 - 21 days after Visit 2, and final study visit (V4) after at maximum 95 days
  Measurement of white blood cells, red blood cells, platelets in blood samples (measurement unit 10^9/L )
Absolute and relative change of hemoglobin | Baseline visit (V1), study visit 2 (V2): 2-4 Weeks after enrolment; Visit 3: 3 - 21 days after Visit 2, and final study visit (V4) after at maximum 95 days
  Measurement in blood samples
Absolute and relative change of hematokrit | Baseline visit (V1), study visit 2 (V2): 2-4 Weeks after enrolment; Visit 3: 3 - 21 days after Visit 2, and final study visit (V4) after at maximum 95 days
  Measurement in blood samples
Absolute and relative change of betahydroxybutyrate level | Baseline visit (V1), study visit 2 (V2): 2-4 Weeks after enrolment; Visit 3: 3 - 21 days after Visit 2, and final study visit (V4) after at maximum 95 days
  Measurement of betahydroxybutyrate level in blood samples for determination of ketosis
Absolute and relative change in blood gas analysis | Baseline visit (V1), study visit 2 (V2): 2-4 Weeks after enrolment; Visit 3: 3 - 21 days after Visit 2, and final study visit (V4) after at maximum 95 days
  Measurement with blood gas analyzer for determination of ketosis
Analysis of the ketonic state with betahydroxybutyrate level | Baseline visit (V1), during 14 days of ketogenic diet or 3 days fasting and final study visit (V4) after at maximum 95 days
  Betahydroxybutyrate measurement from blood samples of the fingertip by patients at home
Analysis of the ketonic state with ketonuria | Baseline visit (V1), during 14 days of ketogenic diet or 3 days fasting and final study visit (V4) after at maximum 95 days
  Ketonuria measured with urine stix by patients at home
Analysis of the ketonic state with acetoacetate in breath | Baseline visit (V1), during 14 days of ketogenic diet or 3 days fasting and final study visit (V4) after at maximum 95 days
  determination of acetoacetate in breath by patients at home
Absolute and relative change of height | Baseline visit (V1), V2 (2-4 Weeks after enrolment); Visit 3 (3 - 21 days after Visit 2 ) and final study visit (V4) after at maximum 95 days
  Determination of height
Absolute and relative change of weight | Baseline visit (V1), V2 (2-4 Weeks after enrolment); Visit 3 (3 - 21 days after Visit 2 ) and final study visit (V4) after at maximum 95 days
  Determination of weight
Absolute and relative change of waist circumference | Baseline visit (V1), V2 (2-4 Weeks after enrolment); Visit 3 (3 - 21 days after Visit 2 ) and final study visit (V4) after at maximum 95 days
  Determination of waist circumference
Relative change of calorimetry | Baseline visit (V1), V2 (2-4 Weeks after enrolment); Visit 3 (3 - 21 days after Visit 2 ) and final study visit (V4) after at maximum 95 days
  Could be determined instead of anthropometric parameters
Changes in Bioimpedance | Baseline visit (V1), V2 (2-4 Weeks after enrolment); Visit 3 (3 - 21 days after Visit 2 ) and final study visit (V4) after at maximum 95 days
  Bioimpedance measurements on each visit
Feeling of hunger, discomforts and problems | In between baseline visit (V1) and final study visit (V4) after at maximum 95 days
  measured and documented at home in a study dietary in between study visits
Acetoacetate-concentrations | In between baseline visit (V1) and final study visit (V4) after at maximum 95 days
  measured and documented at home in a study dietary in between study visits

OTHER OUTCOMES:
Changes of renal functional panel in 24-h-urine | Baseline and during 14 days of ketogenic diet or 3 days fasting
  Urin samples will be collected before and during the dietary intervention for the determination of creatinine, uric acid and urea (measurement unit mg/24h)
Changes of electrolytes and minerals in 24-h-urine | Baseline and during 14 days of ketogenic diet or 3 days fasting
  Urin samples will be collected before and during the dietary intervention for the determination of sodium, natrium, potassium, magnesium, chloride, phosphate (measurement unit mmol/24h )
Changes of glucose in 24-h-urine | Baseline and during 14 days of ketogenic diet or 3 days fasting
  Urin samples will be collected before and during the dietary intervention
Changes of albumin in 24-h-urine | Baseline and during 14 days of ketogenic diet or 3 days fasting
  Urin samples will be collected before and during the dietary intervention
Analysis of stool samples | Baseline and during 14 days of ketogenic diet or 3 days fasting
  Stool samples will be collected before and during the dietary intervention and analysed
Changes of renal functional panel in spot urine | Baseline and during 14 days of ketogenic diet or 3 days fasting
  Urin samples will be collected before and during the dietary intervention for the determination of creatinine, uric acid and urea (measurement unit g/24h)
Changes of electrolytes and minerals in spot urine | Baseline and during 14 days of ketogenic diet or 3 days fasting
  Urin samples will be collected before and during the dietary intervention for the determination of sodium, natrium, potassium, magnesium, chloride, phosphate (measurement unit mmol/24h)
Changes of albumin in spot urine | Baseline and during 14 days of ketogenic diet or 3 days fasting
  Urin samples will be collected before and during the dietary intervention
Changes of glucose in spot urine | Baseline and during 14 days of ketogenic diet or 3 days fasting
  Urin samples will be collected before and during the dietary intervention
Changes in urinary doubly refractile lipid bodies | Baseline and during 14 days of ketogenic diet or 3 days fasting
  Urin samples will be collected before and during the dietary intervention

CONTACTS AND LOCATIONS:
Overall Officials: Roman-Ulrich Müller, Prof., Principal Investigator — Department II of Internal Medicine, University of Cologne
Locations (1):
- Department II of Internal Medicine, University Hospital Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Torres JA, Kruger SL, Broderick C, Amarlkhagva T, Agrawal S, Dodam JR, Mrug M, Lyons LA, Weimbs T. Ketosis Ameliorates Renal Cyst Growth in Polycystic Kidney Disease. Cell Metab. 2019 Dec 3;30(6):1007-1023.e5. doi: 10.1016/j.cmet.2019.09.012. Epub 2019 Oct 17. PMID 31631001